CLINICAL TRIAL: NCT06467318
Title: Does Non-Steroidal Anti-inflammatory Drugs Decrease the Quality of Pleurodesis After Mechanical Pleural Abrasion/Pleurectomy for Treatment of Pneumothorax?
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Bavly Malak, Assistant lecturer in cardio thoracic department, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU MD64/2024
Record Dates: First submitted 2024-06-09; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Primary and Secondary Spontaneous Pneumothorax
MeSH Terms: interventions — Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants post mechanical pleurodesis taking classic pain management with NSAID (Active Comparator)
  Interventions: Drug: NSAID, Paracetamol
- Participants post mechanical pleurodesis taking classic pain management without NSAID (Active Comparator)
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — Participants post mechanical pleurodesis on pneumothorax will be divided into two groups: Group A: patients taking classic pain management with NSAID. Group B: patients taking classic pain management without NSAID.
  Arms: Participants post mechanical pleurodesis taking classic pain management without NSAID
Drug: NSAID, Paracetamol — Participants post mechanical pleurodesis on pneumothorax will be divided into two groups: Group A: patients taking classic pain management with NSAID. Group B: patients taking classic pain management without NSAID.
  Arms: Participants post mechanical pleurodesis taking classic pain management with NSAID

SUMMARY:
Investigators aim to assess if NSAIDs affect the quality of pleurodesis resulting from mechanical pleurodesis (open surgery or VATS) regarding : Primary outcome: Recurrence of pneumothorax in 6 monthes. (assessed by X ray after 2 weeks and 6 months or symptoms requiring X ray at any timing) Secondary outcome: ▪ Adjusted Length of stay ( from day zero surgery day to discharge ). ▪ Time of removal of the chest Tube .(relatively longer with air leak presence). ▪ Need of opioids (N-SAID may decrease the need of opioids) .

DETAILED DESCRIPTION:
Pneumothorax is a relatively common clinical problem which can occur in individuals of any age. Irrespective of aetiology (primary, or secondary to lung disorders or injury), immediate management depends on the extent of cardiorespiratory impairment, degree of symptoms and size of pneumothorax.Non-steroidal anti-inflammatory drugs (NSAIDs) are being used with increasing frequency, due to their potent analgesic effects without having side-effects on the central neural system and additionally due to the large number and varieties of these agents. The analgesic, antiinflammatory properties, and efficacy of NSAIDs in a wide variety of diseases have been already established . Wound healing and formation of adhesions involve inflammation, cell proliferation, matrix deposition, and neovascularization. The exact mechanism by which NSAIDs affect collagen deposition and the time course of the events leading to the formation of fibrin and of adhesions after pleurodesis have not been completely elucidated until now. NSAIDs can inhibit the inflammatory process and the formation of fibrosis, due to their ability to suppress prostaglandin synthesis .

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with primary or secondary spontaneous pneumothorax
* Age: All age groups are included
* Approach: Open and Video assisted thoracoscopic surgery ( Open and VATS pleurodesis).

Exclusion Criteria:

* Refusal of procedure or participation in the study.
* Patient with any contra indication for NSAID (bleeding tendency , CKD , gastritis , allergy to NSAID ,…..)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence of pneumothorax | With in 6 months or earlier with any new symptoms.
  Non-steroidal anti-inflammatory drugs (NSAIDs) are being used with increasing frequency, due to their potent analgesic effects without having side-effects on the central neural system and additionally due to the large number and varieties of these agents. The analgesic, anti inflammatory properties, and efficacy of NSAIDs in a wide variety of diseases have been already established. Wound healing and formation of adhesions involve inflammation, cell proliferation, matrix deposition, and neovascularization. The exact mechanism by which NSAIDs affect collagen deposition and the time course of the events leading to the formation of fibrin and of adhesions after pleurodesis have not been completely elucidated until now. NSAIDs can inhibit the inflammatory process and the formation of fibrosis, due to their ability to suppress prostaglandin synthesis

SECONDARY OUTCOMES:
Measuring adjusted Length of stay | Around 2 weeks
  from day of surgery to discharge (assessed up to 2 weeks )

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided